CLINICAL TRIAL: NCT01754506
Title: Testing Fish Oil Derivatives In Healing Of Chronic Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jodi McDaniel, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011H0228; 1R21NR012803-01A1 (NIH)
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Venous Stasis Ulcers
Keywords: leg ulcers; wounds; fish oil; lipid mediators; chronic venous stasis ulcers
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer; Wounds and Injuries | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA+DHA (Experimental): EPA+DHA (fish oil)
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): mineral oil
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — EPA + DHA Group subjects (n=54) will be given n-3 fatty acid supplement softgels

SUMMARY:
The purpose of this study is to test the efficacy of an oral, nutrient intervention containing the bioactive components of fish oil to promote healing of chronic venous leg ulcers (CVLU). If this systemic, nutrient intervention is found to alter the microenvironment of CVLU, the science of wound healing and care of patients with CVLU will be vastly improved.

DETAILED DESCRIPTION:
The pathogenesis of CVLU involves high numbers of activated polymorphonuclear leukocytes (PMN) that are associated with persistent inflammation in the wound bed 5-9. We propose to test the efficacy of an oral, nutrient intervention containing the bioactive components of fish oil to assuage PMN activity and promote healing of CVLU. If this systemic, nutrient intervention is found to alter the microenvironment of CVLU, the science of wound healing and care of patients with CVLU will be vastly improved.

The purpose of this study is to test three fundamental corollaries of our organizing hypothesis in a 2-group, double-blind, randomized, experimental design on CVLU patients. The findings from the proposed experiments will increase our understanding of lipid mediators that influence wound healing and PMN function, and may lead to an innovative approach to reduce the physical and emotional burdens of nonhealing or recurrent CVLU.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* ages 18-85 years
* having at least one existing CVLU between the ankle and knee for ≥ 3 months
* medical clearance to take 81mg/d of aspirin
* prescribed compression therapy; ambulatory
* ankle brachial pressure index (ABPI) of ≥ 0.8
* target wound of ≥ 1 x 1 inches (6.25 cm2)
* can understand English and sign own consent

Exclusion Criteria:

* allergy to fish or seafood
* exposed bone, tendon or fascia around target wound
* receiving warfarin or Plavix therapy
* immunologic related condition (e.g. Crohn's disease, systemic lupus erythematosus)
* chronic inflammatory skin diseases (e.g. pyoderma gangrenosum, psoriasis)
* requiring non-steroidal anti-inflammatory drugs > 2x a week
* nutritional supplements or corticosteroids
* chronic renal insufficiency
* already in a study related to CVLU.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Levels of eicosapentaenoic (EPA)+ docosahexaenoic (DHA)-derived lipid mediators and proinflammatory cytokines in blood and CVLU wound fluid | 0, 28, 56 days

SECONDARY OUTCOMES:
PMN counts and levels of PMN-derived proteases in CVLU wound fluid | 0, 28, 56 days

OTHER OUTCOMES:
Re-epithelialization | 28, 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Jodi C McDaniel, PhD, RN, Principal Investigator — The Ohio State University College of Nursing
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

REFERENCES:
- [Derived] McDaniel JC. Dietary supplement use by older adults with chronic venous leg ulcers: A retrospective, descriptive study. Wound Repair Regen. 2020 Jul;28(4):561-572. doi: 10.1111/wrr.12821. Epub 2020 May 4. PMID 32319144